CLINICAL TRIAL: NCT03761784
Title: A Phase 3 Multi-Center, Double-Blind, Randomized, Vehicle-Controlled Study of S6G5T-3 in the Treatment of Acne Vulgaris
Brief Title: A Study of S6G5T-3 in the Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sol-Gel Technologies, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SGT-65-04
Record Dates: First submitted 2018-11-30; First posted 2018-12-03 (Actual); Results first posted 2021-12-01 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Acne Vulgaris
Keywords: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- S6G5T-3 (Experimental): Participants will topically apply S6G5T-3 cream, once daily to face for 12 weeks.
  Interventions: Drug: S6G5T-3
- S6G5T-8 Vehicle Cream (Placebo Comparator): Participants will topically apply S6G5T-8 vehicle cream, once daily to face for 12 weeks.
  Interventions: Drug: S6G5T-8

INTERVENTIONS:
Drug: S6G5T-3 — Once a day topical cream
  Other Names: Encapsulated Benzoyl Peroxide (E-BPO) and Encapsulated Tretinoin (E-ATRA) Cream, (E-BPO/E-ATRA Cream)
  Arms: S6G5T-3
Drug: S6G5T-8 — Once a day topical cream
  Other Names: Vehicle
  Arms: S6G5T-8 Vehicle Cream

SUMMARY:
To assess the efficacy of S6G5T-3 compared to its Vehicle when applied once daily for 12 weeks in participants with acne vulgaris.

DETAILED DESCRIPTION:
In this Phase 3, multi-center, double-blind, randomized, vehicle-controlled, parallel-group pivotal study, participants will be admitted only after a written informed consent has been obtained and after all inclusion/exclusion criteria have been met. Male and female participants at least 9 years of age with facial acne vulgaris will be eligible for enrollment for daily treatment with S6G5T-3 or its vehicle S6G5T-8, for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must sign an Institutional Review Board (IRB) approved written informed consent for this study.
2. Male and female 9 years of age and older.
3. Have 2 or fewer cysts or nodules.

Exclusion Criteria:

1. More than 2 acne nodules or cysts (defined as an inflammatory lesion greater than or equal to 5 millimeter (mm) in diameter).
2. Acne conglobata, acne fulminans, and secondary acne (for example, chloracne, drug-induced acne).
3. History of blood dyscrasia (for example, leukemia, haemophilia, sickle cell anemia, multiple myeloma).
4. Underlying disease that requires the use of interfering topical or systemic therapy.
5. Other dermatological conditions that require the use of interfering topical or systemic therapy or that might interfere with study assessments such as, but not limited to, atopic dermatitis, perioral dermatitis, or rosacea.

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 424 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology Consulting Services, High Point, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to receive either S6G5T-3 (Encapsulated Benzoyl Peroxide [E-BPO] and Encapsulated Tretinoin [E-ATRA] Cream, 3%/0.1% [E-BPO/E-ATRA Cream, 3%/0.1%]) or vehicle in a 2:1 ratio.
Groups:
- S6G5T-3: Participants topically applied S6G5T-3, once daily to face for 12 weeks.
- S6G5T-8 Vehicle Cream: Participants topically applied S6G5T-8 vehicle cream, once daily to face for 12 weeks.
Period: Overall Study
Arm/Group | S6G5T-3 | S6G5T-8 Vehicle Cream
Started | 281 | 143
Received at Least 1 Dose of Study Drug | 274 | 139
Completed | 249 | 131
Not Completed | 32 | 12
Not completed — Adverse Event | 4 | 0
Not completed — Lost to Follow-up | 10 | 7
Not completed — Pregnancy | 1 | 0
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Parent or Guardian | 4 | 1
Not completed — Withdrawal by Subject | 9 | 4
Not completed — Physician Decision | 1 | 0
Not completed — Other Than Specified | 1 | 0

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population consisted of all randomized participants who were dispensed study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | S6G5T-3 | S6G5T-8 Vehicle Cream | Total
Number analyzed (Participants) | 281 | 143 | 424
Age, Continuous [Mean (Standard Deviation); unit: Years] | 20.9 (8.48) | 21.4 (8.62) | 21.1 (8.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 175 | 83 | 258
  Male | 106 | 60 | 166
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 102 | 44 | 146
  Not Hispanic or Latino | 178 | 98 | 276
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 26 | 10 | 36
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 53 | 20 | 73
  White | 194 | 109 | 303
  More than one race | 6 | 1 | 7
  Unknown or Not Reported | 0 | 0 | 0
Baseline Acne Lesion Count on the Face [Mean (Standard Deviation); unit: Lesions] — Inflammatory lesions were characterized by papules, pustules, nodules, and cysts. Non-inflammatory lesions were characterized by open comedones (blackheads) and closed comedones (whiteheads).
  Lesions
    Inflammatory Lesions | 33.5 (14.62) | 33.5 (14.69) | 33.5 (14.63)
    Non-Inflammatory lesions | 48.6 (20.24) | 47.1 (19.97) | 48.1 (20.14)
Baseline Investigator's Global Assessment (IGA) [Count of Participants; unit: Participants] — Investigator's Global Assessment (IGA), where Investigator's rated the participant's acne from 0 (Clear) to 4 (Severe). A higher score indicated an increase in severity of facial acne.
  Participants
    0 - Clear | 0 | 0 | 0
    1 - Almost Clear | 0 | 0 | 0
    2 - Mild | 0 | 0 | 0
    3 - Moderate | 251 | 132 | 383
    4 - Severe | 30 | 11 | 41

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving an IGA Score of Clear or Almost Clear and a Score ≥2 Grades Less Than Baseline
Description: Percentage of participants in each treatment group achieving an acne severity IGA score of "clear (score=0)" or "almost clear (score=1)" and achieving an acne severity IGA score of at least 2 grades less than Baseline.
Time Frame: Baseline through Week 12
Population: The ITT population consisted of all randomized participants who were dispensed study drug. Multiple imputation (MCMC) was used to impute missing values.
Measure: Number; unit: percentage of participants
Arm/Group | S6G5T-3 | S6G5T-8 Vehicle Cream
Number analyzed (Participants) | 281 | 143
percentage of participants | 38.5 | 11.5

2. Primary Outcome: Change From Baseline in Inflammatory Lesion Counts on the Face at Week 12
Description: Inflammatory lesions were characterized by papules, pustules, nodules, and cysts. Least squares means and standard deviations from an analysis of covariance (ANCOVA) with factors of treatment group and analysis center and the respective Baseline lesion count as a covariate. For the inflammatory lesion count analysis, the interaction of treatment by analysis center was included in the model based on the conclusion from the pooling analysis. Negative least squares means values represent decrease from Baseline.
Time Frame: Baseline, Week 12
Population: The ITT population consisted of all randomized participants who were dispensed study drug. MCMC was used to impute missing values.
Measure: Least Squares Mean (Standard Deviation); unit: Inflammatory Lesions
Arm/Group | S6G5T-3 | S6G5T-8 Vehicle Cream
Number analyzed (Participants) | 281 | 143
Inflammatory Lesions | -21.6 (10.67) | -14.8 (11.03)

3. Primary Outcome: Change From Baseline in Non-Inflammatory Lesion Counts on the Face at Week 12
Description: Non-inflammatory lesions were characterized by open comedones (blackheads) and closed comedones (whiteheads). Least squares means and standard deviations from an ANCOVA with factors of treatment group and analysis center and the respective Baseline lesion count as a covariate. Negative least squares means values represent decrease from Baseline.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Deviation); unit: Non-Inflammatory Lesions
Arm/Group | S6G5T-3 | S6G5T-8 Vehicle Cream
Number analyzed (Participants) | 281 | 143
Non-Inflammatory Lesions | -29.7 (15.26) | -19.8 (15.84)

4. Secondary Outcome: Percent Change From Baseline in Non-Inflammatory Lesion Counts on the Face at Week 12
Description: as for outcome 3
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Deviation); unit: Percent Change
Arm/Group | S6G5T-3 | S6G5T-8 Vehicle Cream
Number analyzed (Participants) | 281 | 143
Percent Change | -61.6 (31.38) | -40.9 (32.63)

5. Secondary Outcome: Percent Change From Baseline in Inflammatory Lesion Counts on the Face at Week 12
Description: Inflammatory lesions were characterized by papules, pustules, nodules, and cysts. Least squares means and standard deviations from an ANCOVA with factors of treatment group and analysis center and the respective Baseline lesion count as a covariate. For the inflammatory lesion count analysis, the interaction of treatment by analysis center was included in the model based on the conclusion from the pooling analysis. Negative least squares means values represent decrease from Baseline.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Deviation); unit: Percent Change
Arm/Group | S6G5T-3 | S6G5T-8 Vehicle Cream
Number analyzed (Participants) | 281 | 143
Percent Change | -66.1 (32.28) | -43.5 (32.87)

6. Secondary Outcome: Percentage of Participants Achieving at Least a 4-Point Reduction on Item 1 (Pimple) of the Patient-Reported Evaluation of Facial Acne (Pre-Face)
Description: Percent of participants in each treatment group achieving at least a 4-point reduction on Item 1 (Pimple) of patient-reported evaluation of facial acne compared to Baseline. The Pre-Face is a 7-item questionnaire that assesses acne vulgaris-related signs, symptoms, and impacts. Item 1 of the questionnaire was to assess the pimples on the participant's face at their worst, in the 24 hours prior to administration on an 11-point numeric rating scale (NRS) ranging from 0 ("no pimples at all") to 10 ("pimples as bad as you can imagine").
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | S6G5T-3 | S6G5T-8 Vehicle Cream
Number analyzed (Participants) | 281 | 143
percentage of participants | 38.9 | 18.6

7. Secondary Outcome: Percentage of Participants Achieving at Least a 4-Point Reduction on Item 5 (Embarrassment) of the Pre-Face
Description: Percent of participants in each treatment group achieving at least a 4-point reduction on Item 5 (Embarrassment) of the patient-reported evaluation of facial acne compared to Baseline. The Pre-Face is a 7-item questionnaire that assesses acne vulgaris-related signs, symptoms, and impacts. Item 5 of the questionnaire was to assess how embarrassed the participant felt because of the acne at their worst in the 24 hours prior to administration on an 11-point NRS ranging from 0 ("not embarrassed at all") to 10 ("extremely embarrassed").
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | S6G5T-3 | S6G5T-8 Vehicle Cream
Number analyzed (Participants) | 281 | 143
percentage of participants | 42.8 | 32.7

8. Secondary Outcome: Change From Baseline in Non-Inflammatory Lesion Counts on the Face at Week 8
Description: as for outcome 3
Time Frame: Baseline, Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Deviation); unit: Non-Inflammatory Lesions
Arm/Group | S6G5T-3 | S6G5T-8 Vehicle Cream
Number analyzed (Participants) | 281 | 143
Non-Inflammatory Lesions | -24.4 (16.44) | -16.9 (15.60)

9. Secondary Outcome: Change From Baseline in Inflammatory Lesion Counts on the Face at Week 8
Description: as for outcome 5
Time Frame: Baseline, Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Deviation); unit: Inflammatory Lesions
Arm/Group | S6G5T-3 | S6G5T-8 Vehicle Cream
Number analyzed (Participants) | 281 | 143
Inflammatory Lesions | -17.2 (12.10) | -12.5 (11.61)

10. Secondary Outcome: Change From Baseline in Non-Inflammatory Lesion Counts on the Face at Week 4
Description: as for outcome 3
Time Frame: Baseline, Week 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Deviation); unit: Non-Inflammatory Lesions
Arm/Group | S6G5T-3 | S6G5T-8 Vehicle Cream
Number analyzed (Participants) | 281 | 143
Non-Inflammatory Lesions | -18.5 (14.16) | -13.4 (13.99)

11. Secondary Outcome: Change From Baseline in Inflammatory Lesion Counts on the Face at Week 4
Description: as for outcome 5
Time Frame: Baseline, Week 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Deviation); unit: Inflammatory Lesions
Arm/Group | S6G5T-3 | S6G5T-8 Vehicle Cream
Number analyzed (Participants) | 281 | 143
Inflammatory Lesions | -13.5 (10.32) | -9.8 (10.28)

ADVERSE EVENTS:
Time Frame: Baseline (Day 0) through end of study (Week 12)
Description: Safety population included randomized participants who were presumed to have used the study drug at least once and who provided at least 1 post-baseline safety evaluation.
Arm/Group | S6G5T-3 | S6G5T-8 Vehicle Cream
All-Cause Mortality (participants affected / at risk) | 0/274 | 0/139
Serious Adverse Events (participants affected / at risk) | 0/274 | 0/139
Other Adverse Events (participants affected / at risk) | 69/274 | 8/139
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | S6G5T-3 (N=274) | S6G5T-8 Vehicle Cream (N=139)
Application site pain (General disorders) | 33 | 0
Application site dryness (General disorders) | 17 | 1
Application site erythema (General disorders) | 14 | 0
Application site exfoliation (General disorders) | 14 | 0
Application site dermatitis (General disorders) | 4 | 1
Application site irritation (General disorders) | 4 | 0
Upper respiratory tract infection (Infections and infestations) | 6 | 3
Headache (Nervous system disorders) | 3 | 1
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the Principal Investigator is not permitted to discuss or publish trial results without Sponsor approval.

DOCUMENTS (2):
  • Study Protocol (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/84/NCT03761784/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-26): https://cdn.clinicaltrials.gov/large-docs/84/NCT03761784/SAP_001.pdf